CLINICAL TRIAL: NCT03325062
Title: Movement Pattern Biofeedback Training After Total Knee Arthroplasty
Acronym: MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of California, San Francisco (Other); University of Delaware (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-1701; R01AG056585 (NIH)
Record Dates: First submitted 2017-10-18; First posted 2017-10-30 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Total Knee Arthroplasty; Older Adults

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are only informed that they will participate in one of two post-operative rehabilitation programs (without specific details). Outcome assessors are also blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: MOVE (Experimental): Movement pattern training in addition to contemporary progressive rehabilitation
  Interventions: Behavioral: Experimental: MOVE
- CONTROL (Active Comparator): Contemporary progressive rehabilitation
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Control — The contemporary progressive rehabilitation program consists of progressive resistive exercise to key lower extremity muscle groups, knee range of motion exercise, weight-bearing exercise, as well as education on symptom management strategies.
  Arms: CONTROL
Behavioral: Experimental: MOVE — The MOVE program emphasizes movement pattern retraining in conjunction with contemporary rehabilitation. More specifically, the MOVE program promotes symmetry in functional knee motion and loading without postural compensation. Intervention uses pressure-sensing shoe insoles to deliver real-time visual biofeedback during activity performance.
  Arms: Experimental: MOVE

SUMMARY:
This research study explores the effects of movement pattern training using real-time biofeedback insoles after total knee arthroplasty. The purpose of this research study is to determine if the addition of a novel movement pattern training program (MOVE) to contemporary progressive rehabilitation leads to improved movement quality and physical function compared to contemporary progressive rehabilitation (CONTROL) alone.

DETAILED DESCRIPTION:
Currently in the United States, more than 700,000 total knee arthroplasty (TKA) surgeries are performed annually, with projections of 3.5 million performed annually by 2030. The increasing incidence of TKA comes with an immediate need for establishing optimal rehabilitation guidelines to remediate common post-TKA physical impairments and improve functional outcomes. Over the past decade, a primary focus of the investigators' TKA rehabilitation research has been on progressive strengthening, which improves muscle strength and physical function, and is now the contemporary approach to TKA rehabilitation. However, a major issue remaining for patients rehabilitating from unilateral TKA is the persistence of atypical movement patterns. These atypical movement patterns, observed during walking and other functional tasks, are characterized by disuse of the surgical limb, resulting in smaller knee extension moments on the surgical limb compared to the non-surgical limb. As a result, atypical movement patterns following unilateral TKA are associated with persistent quadriceps weakness and poor physical function.

The investigators will conduct a randomized controlled trial of 150 participants undergoing unilateral TKA to determine if the addition of a novel movement pattern training program (MOVE) to contemporary, progressive rehabilitation improves movement pattern quality more than contemporary progressive rehabilitation alone (CONTROL). The secondary goal is to determine if movement pattern training improves long-term physical function. Testing will occur pre-operatively and after TKA at 10 weeks (end of intervention), 6 months (primary endpoint), and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. 50-85 years old
2. primary, unilateral knee arthroplasty for end-stage osteoarthritis

Exclusion Criteria:

1. Moderate to severe contralateral knee OA (>4/10 on verbal pain rating (VPR) or KL grade >3)
2. Current smoker
3. Drug abuse
4. Comorbid conditions that substantially limit physical function or would interfere with the participant's ability to successfully complete rehabilitation (e.g. neurologic, vascular, cardiac problems, or ongoing medical treatments)
5. Discharge to location other than home after surgery
6. Unstable orthopedic conditions that limit function
7. Uncontrolled diabetes (hemoglobin A1c level >8.0)
8. Body mass index >40 kg/m2
9. Surgical complication necessitating an altered course of rehabilitation
10. Previous contralateral TKA
11. Unable to safely walk 30m without an assistive device

Exclusion criteria for MRI

1. Ferromagnetic metal implants or pacemakers
2. Other contraindications to MRI

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Change in Peak Knee Extension Moment (PKEM) during walking at fixed speed | Baseline, 10 weeks, 6 months, and 2 years after surgery
  Peak Knee Extension Moment (PKEM) during walking at a fixed speed of 1.0 m/s

SECONDARY OUTCOMES:
Change in PKEM during activities | Baseline, 10 weeks, 6 months, and 2 years after surgery
  PKEM during walking at self-selected gait speed, rising and lowering from a chair, and stepping up and down a step
Change in Six-minute Walk (6MW) Test | Baseline, 10 weeks, 6 months, and 2 years after surgery
  Developed and used extensively to measure endurance, measures the distance walked in six minutes.
Change in Stair Climbing Test (SCT) | Baseline, 10 weeks, 6 months, and 2 years after surgery
  Measures a higher level of function that minimizes the possibility of a ceiling effect
Change in 30-Second Sit-to-Stand Test (30-STS) | Baseline, 10 weeks, 6 months, and 2 years after surgery
  Assesses lower body strength and the fatigue effect caused by the number of sit-to-stand repetitions.
Change in Accelerometer-based Physical Activity | Baseline, 10 weeks, 6 months, and 2 years after surgery
  Assesses daily physical activity levels and number of steps.
Change in Quadriceps Strength | Baseline, 10 weeks, 6 months, and 2 years after surgery
  Assesses the maximal voluntary isometric contraction strength of the quadriceps muscle
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 10 weeks, 6 months, and 2 years after surgery
  Assesses self-reported physical function. Scale assess pain, stiffness, and physical function in patients with hip and / or knee osteoarthritis. Total score range is 0-96. Total score is computed by summing three subscales: pain (range 0-20), stiffness (range 0-8), and functional limitations (range 0-68), then dividing by total points possible. Higher scores indicate worse pain, stiffness, and functional limitations.
Change in Veterans RAND 12 item health survey (VR-12) | Baseline, 10 weeks, 6 months, and 2 years after surgery
  A generic instrument to measure health related quality of life. The VR-12 has two subscales, the Physical Component Score (PCS) and the Mental Component Score (MCS). The PCS and MCS summary scores are standardized using a t-score transformation and normed to a U.S. population (based on a 1990 norm) of a score of 50 and a standard deviation of 10.
Change in Timed Up and Go (TUG) | Baseline, 10 weeks, 6 months, and 2 years after surgery
  The TUG evaluates mobility through the time required to rise from an arm chair, walk 3 meters, turn and walk back to the arm chair, and return to a seated position.
Change in knee range of motion (ROM) | Baseline, 10 weeks, 6 months, and 2 years after surgery
  Assesses the mobility of the knee joint.
Adherence to the intervention | 10 weeks after surgery
  Assesses the adherence of subjects as measured by home exercise program logs and number of clinical sessions attended.
Satisfaction with rehabilitation program | 10 weeks after surgery
  Assesses the satisfaction of subjects with their assigned rehabilitation program using a 5-point Likert scale ranging from "very unsatisfied" to "very satisfied".

OTHER OUTCOMES:
Change in contralateral knee whole-organ MRI scoring method (WORMS) total sum score | 10 weeks and 2 years after surgery
  Whole-organ MRI scoring method (WORMS) is a semi-quantitative, MRI-based scoring system that evaluates the integrity of articular cartilage, ligaments/tendons, menisci, bone marrow lesions, effusion, subchondral cysts, loose bodies, and popliteal cysts. The Total sum score ranges from 0-129 and is computed by summing the following subscales: Cartilage (0-36), Ligaments/tendons (0-24), Meniscus (0-24), Bone marrow Lesions (0-18), Joint Effusion (0-3), Subchondral Cysts (0-18), Loose Bodies (0-3), and Popliteal Cyst (0-3). Higher scores indicate greater amounts of joint degeneration.
Incidence of contralateral TKA | 2 years after surgery
  Number of participants who have a contralateral TKA

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Stevens-Lapsley, PT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be shared in a publication, which will be available through pubmed within a year of publication.
Supporting Information: ICF, CSR
Time Frame: Publications will be made available to the public through PubMed Central within one year after the date of publication.

REFERENCES:
- [Background] Christiansen CL, Bade MJ, Davidson BS, Dayton MR, Stevens-Lapsley JE. Effects of Weight-Bearing Biofeedback Training on Functional Movement Patterns Following Total Knee Arthroplasty: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2015 Sep;45(9):647-55. doi: 10.2519/jospt.2015.5593. Epub 2015 Jul 24. PMID 26207975
- [Background] Zeni J Jr, Abujaber S, Flowers P, Pozzi F, Snyder-Mackler L. Biofeedback to promote movement symmetry after total knee arthroplasty: a feasibility study. J Orthop Sports Phys Ther. 2013 Oct;43(10):715-26. doi: 10.2519/jospt.2013.4657. Epub 2013 Aug 30. PMID 23892267
- [Background] McClelland J, Zeni J, Haley RM, Snyder-Mackler L. Functional and biomechanical outcomes after using biofeedback for retraining symmetrical movement patterns after total knee arthroplasty: a case report. J Orthop Sports Phys Ther. 2012 Feb;42(2):135-44. doi: 10.2519/jospt.2012.3773. Epub 2012 Feb 1. PMID 22333656